CLINICAL TRIAL: NCT04050956
Title: French Cohort of Myocardial Infarction Evaluation
Acronym: FRENCHIE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: NI17011
Record Dates: First submitted 2019-08-02; First posted 2019-08-09 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Registry; Outcomes; Medico-economic evaluation; Comorbidities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocardial infarction: As it is an observational study, no intervention is planned. However, nested clinical interventional trials are planned for which a specific registration will be done

SUMMARY:
Over the last two decades, considerable progress has been made in the management of Acute Myocardial Infarction (AMI), both in the acute phase and in monitoring beyond the hospital phase. Nevertheless, the evolution of care practices and their impact on the mid- and long-term prognosis of patients admitted to the intensive care unit for acute myocardial infarction remain relatively little studied exhaustively.

The aim of this study is to assess the profile of AMI patients, their management and follow-up in order to evaluate the relationship between these factors and outcomes.

DETAILED DESCRIPTION:
The FRENCHIE registry is a French multicenter prospective observational study. All the eligible consecutive patients admitted within 48 hours after symptom onset in a cardiac ICU for an acute myocardial infarction.

This hospital registry will be linked to the national databases, in order to collect follow-up clinical outcomes and health care consumption.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction (MI) within 48h of symptom onset, characterized by the typical increased or fall of troponin (or CPKMB) associated with at least one of the following elements :
* Symptoms compatible with myocardial ischemia
* Appearance of pathological Q waves
* ST- T changes compatible with myocardial ischemia (ST segment elevation or depression, T-wave inversion)
* Written consent.
* Covered by French medical insurance ("Sécurité Sociale")

Exclusion Criteria:

* Iatrogenic MI defined as MI occurring within 48h of a therapeutic procedure
* AMI diagnosis invalidated in favor of another diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive eligible (cf eligibility criteria) patients admitted in one of the Intensive Coronary Units participating to the study.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2029-03-22 (Estimated); Study Completion 2049-03-22 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Through the end of initial hospitalization, an average of 5 days
  In-hospital mortality
In-hospital outcomes | Through the end of initial hospitalization, an average of 5 days
  To measure the in-hospital major cardiovascular events : recurrence of AMI, myocardial revascularization, stroke
Lipopretein 1 evolution | 9 months after the end of initial hospitalization
  To evaluate plasma concentrations of Lpa and its dynamic pattern during hospital index and 3-9 months following hospitalization.

SECONDARY OUTCOMES:
Cardiovascular outcomes during follow-up | Up to 20 years
  All cause death and Cardiovascular events including non fatal Myocardial Infarction, non fatal stroke, revascularization, hospitalization for other cardiovascular causes including Bleeding leading to hospitalization
Non cardiovascular outcomes during follow-up | Up to 20 years
  All cause death and Non-cardiovascular events leading to to hospitalizations
Relationship between patients profile and mortality and cardiovascular morbidity outcomes according to management | Up to 20 years
  All cause death and cardiovascular events including non fatal MI, non fatal stroke, revascularization, hospitalization for other cardiovascular causes including Bleeding leading to hospitalization according to patient's management
Relationship between patients profile and mortality and non-cardiovascular morbidity outcomes according to management | Up to 20 years
  All cause death and Non-cardiovascular events leading to to hospitalizations according to patient's management
Oral comorbidities | Up to 20 years
  Prevalence of oral pathology and its relationship with early, mid, and long-term prognosis and outcomes
Sleep disordered breathing comorbidities | Up to 20 years
  To assess the prevalence of sleep disordered breathing comorbidities and the relationship with early, mid, and long-term prognosis and outcomes
Evaluate the path of care combined with patient care practices following an acute myocardial infarction | Up to 20 years
  Evaluate the path of care and patient care practices following an acute myocardial infarction : Reimbursed or prescribed treatments, combined with number of visits, biological and tests performed
Evaluate the relevance of European Society of Cardiology (ESC), American Heart Association/American College of Cardiology (AHA / ACC) guidelines regarding management of AMI patients | Up to 20 years
  Evaluate the relevance of ESC, AHA/ACC guidelines regarding management of AMI patients
Cost-utility: incremental (or decremental) cost-utility ratio during follow-up | Up to 20 years
  Medical care costs for the index hospitalization and during follow-up period are assessed using a combination of resource-based and event-based methods. In-hospital resource utilization are based on diagnosis and procedural codes and length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gabriel STEG, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hasdai D, Behar S, Wallentin L, Danchin N, Gitt AK, Boersma E, Fioretti PM, Simoons ML, Battler A. A prospective survey of the characteristics, treatments and outcomes of patients with acute coronary syndromes in Europe and the Mediterranean basin; the Euro Heart Survey of Acute Coronary Syndromes (Euro Heart Survey ACS). Eur Heart J. 2002 Aug;23(15):1190-201. doi: 10.1053/euhj.2002.3193. PMID 12127921
- [Background] Pedersen TR, Kjekshus J, Berg K, Haghfelt T, Faergeman O, Faergeman G, Pyorala K, Miettinen T, Wilhelmsen L, Olsson AG, Wedel H; Scandinavian Simvastatin Survival Study Group. Randomised trial of cholesterol lowering in 4444 patients with coronary heart disease: the Scandinavian Simvastatin Survival Study (4S). 1994. Atheroscler Suppl. 2004 Oct;5(3):81-7. doi: 10.1016/j.atherosclerosissup.2004.08.027. No abstract available. PMID 15531279
- [Background] Sacks FM, Pfeffer MA, Moye LA, Rouleau JL, Rutherford JD, Cole TG, Brown L, Warnica JW, Arnold JM, Wun CC, Davis BR, Braunwald E. The effect of pravastatin on coronary events after myocardial infarction in patients with average cholesterol levels. Cholesterol and Recurrent Events Trial investigators. N Engl J Med. 1996 Oct 3;335(14):1001-9. doi: 10.1056/NEJM199610033351401. PMID 8801446
- [Background] Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol lowering with simvastatin in 20,536 high-risk individuals: a randomised placebo-controlled trial. Lancet. 2002 Jul 6;360(9326):7-22. doi: 10.1016/S0140-6736(02)09327-3. PMID 12114036
- [Background] GUSTO investigators. An international randomized trial comparing four thrombolytic strategies for acute myocardial infarction. N Engl J Med. 1993 Sep 2;329(10):673-82. doi: 10.1056/NEJM199309023291001. PMID 8204123
- [Background] Andersen HR, Nielsen TT, Rasmussen K, Thuesen L, Kelbaek H, Thayssen P, Abildgaard U, Pedersen F, Madsen JK, Grande P, Villadsen AB, Krusell LR, Haghfelt T, Lomholt P, Husted SE, Vigholt E, Kjaergard HK, Mortensen LS; DANAMI-2 Investigators. A comparison of coronary angioplasty with fibrinolytic therapy in acute myocardial infarction. N Engl J Med. 2003 Aug 21;349(8):733-42. doi: 10.1056/NEJMoa025142. PMID 12930925
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Danchin N, Vaur L, Genes N, Etienne S, Angioi M, Ferrieres J, Cambou JP. Treatment of acute myocardial infarction by primary coronary angioplasty or intravenous thrombolysis in the "real world": one-year results from a nationwide French survey. Circulation. 1999 May 25;99(20):2639-44. doi: 10.1161/01.cir.99.20.2639. PMID 10338456
- [Background] Danchin N, Vaur L, Genes N, Renault M, Ferrieres J, Etienne S, Cambou JP. Management of acute myocardial infarction in intensive care units in 1995: a nationwide French survey of practice and early hospital results. J Am Coll Cardiol. 1997 Dec;30(7):1598-605. doi: 10.1016/s0735-1097(97)00371-9. PMID 9385882
- [Background] Hanania G, Cambou JP, Gueret P, Vaur L, Blanchard D, Lablanche JM, Boutalbi Y, Humbert R, Clerson P, Genes N, Danchin N; USIC 2000 Investigators. Management and in-hospital outcome of patients with acute myocardial infarction admitted to intensive care units at the turn of the century: results from the French nationwide USIC 2000 registry. Heart. 2004 Dec;90(12):1404-10. doi: 10.1136/hrt.2003.025460. PMID 15547013
- [Background] Danchin N, Blanchard D, Steg PG, Sauval P, Hanania G, Goldstein P, Cambou JP, Gueret P, Vaur L, Boutalbi Y, Genes N, Lablanche JM; USIC 2000 Investigators. Impact of prehospital thrombolysis for acute myocardial infarction on 1-year outcome: results from the French Nationwide USIC 2000 Registry. Circulation. 2004 Oct 5;110(14):1909-15. doi: 10.1161/01.CIR.0000143144.82338.36. Epub 2004 Sep 27. PMID 15451803
- [Background] Ferrieres J, Cambou JP, Gueret P, Boutalbi Y, Lablanche JM, Hanania G, Genes N, Cantet C, Danchin N. Effect of early initiation of statins on survival in patients with acute myocardial infarction (the USIC 2000 Registry). Am J Cardiol. 2005 Feb 15;95(4):486-9. doi: 10.1016/j.amjcard.2004.10.016. PMID 15695134
- [Background] Heidenreich PA, Alloggiamento T, Melsop K, McDonald KM, Go AS, Hlatky MA. The prognostic value of troponin in patients with non-ST elevation acute coronary syndromes: a meta-analysis. J Am Coll Cardiol. 2001 Aug;38(2):478-85. doi: 10.1016/s0735-1097(01)01388-2. PMID 11499741
- [Background] Cambou JP, Simon T, Mulak G, Bataille V, Danchin N. The French registry of Acute ST elevation or non-ST-elevation Myocardial Infarction (FAST-MI): study design and baseline characteristics. Arch Mal Coeur Vaiss. 2007 Jun-Jul;100(6-7):524-34. PMID 17893635
- [Background] Hanssen M, Cottin Y, Khalife K, Hammer L, Goldstein P, Puymirat E, Mulak G, Drouet E, Pace B, Schultz E, Bataille V, Ferrieres J, Simon T, Danchin N; FAST-MI 2010 Investigators. French Registry on Acute ST-elevation and non ST-elevation Myocardial Infarction 2010. FAST-MI 2010. Heart. 2012 May;98(9):699-705. doi: 10.1136/heartjnl-2012-301700. PMID 22523054
- [Background] Danchin N, Coste P, Ferrieres J, Steg PG, Cottin Y, Blanchard D, Belle L, Ritz B, Kirkorian G, Angioi M, Sans P, Charbonnier B, Eltchaninoff H, Gueret P, Khalife K, Asseman P, Puel J, Goldstein P, Cambou JP, Simon T; FAST-MI Investigators. Comparison of thrombolysis followed by broad use of percutaneous coronary intervention with primary percutaneous coronary intervention for ST-segment-elevation acute myocardial infarction: data from the french registry on acute ST-elevation myocardial infarction (FAST-MI). Circulation. 2008 Jul 15;118(3):268-76. doi: 10.1161/CIRCULATIONAHA.107.762765. Epub 2008 Jun 30. PMID 18591434
- [Background] Danchin N, Puymirat E, Steg PG, Goldstein P, Schiele F, Belle L, Cottin Y, Fajadet J, Khalife K, Coste P, Ferrieres J, Simon T; FAST-MI 2005 Investigators. Five-year survival in patients with ST-segment-elevation myocardial infarction according to modalities of reperfusion therapy: the French Registry on Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) 2005 Cohort. Circulation. 2014 Apr 22;129(16):1629-36. doi: 10.1161/CIRCULATIONAHA.113.005874. Epub 2014 Mar 21. PMID 24657993
- [Background] Ferrieres J, Bataille V, Leclercq F, Geslin P, Ruidavets JB, Grollier G, Bernard P, Cambou JP, Simon T, Danchin N. Patterns of statin prescription in acute myocardial infarction: the French registry of Acute ST-elevation or non-ST-elevation Myocardial Infarction (FAST-MI). Atherosclerosis. 2009 Jun;204(2):491-6. doi: 10.1016/j.atherosclerosis.2008.09.031. Epub 2008 Oct 8. PMID 19004441
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Puymirat E, Simon T, Steg PG, Schiele F, Gueret P, Blanchard D, Khalife K, Goldstein P, Cattan S, Vaur L, Cambou JP, Ferrieres J, Danchin N; USIK USIC 2000 Investigators; FAST MI Investigators. Association of changes in clinical characteristics and management with improvement in survival among patients with ST-elevation myocardial infarction. JAMA. 2012 Sep 12;308(10):998-1006. doi: 10.1001/2012.jama.11348. PMID 22928184
- [Background] Puymirat E, Schiele F, Steg PG, Blanchard D, Isorni MA, Silvain J, Goldstein P, Gueret P, Mulak G, Berard L, Bataille V, Cattan S, Ferrieres J, Simon T, Danchin N; FAST-MI investigators. Determinants of improved one-year survival in non-ST-segment elevation myocardial infarction patients: insights from the French FAST-MI program over 15 years. Int J Cardiol. 2014 Nov 15;177(1):281-6. doi: 10.1016/j.ijcard.2014.09.023. Epub 2014 Sep 28. PMID 25499393
- [Background] Puymirat E, Taldir G, Aissaoui N, Lemesle G, Lorgis L, Cuisset T, Bourlard P, Maillier B, Ducrocq G, Ferrieres J, Simon T, Danchin N. Use of invasive strategy in non-ST-segment elevation myocardial infarction is a major determinant of improved long-term survival: FAST-MI (French Registry of Acute Coronary Syndrome). JACC Cardiovasc Interv. 2012 Sep;5(9):893-902. doi: 10.1016/j.jcin.2012.05.008. PMID 22995875
- [Background] Franklin K, Goldberg RJ, Spencer F, Klein W, Budaj A, Brieger D, Marre M, Steg PG, Gowda N, Gore JM; GRACE Investigators. Implications of diabetes in patients with acute coronary syndromes. The Global Registry of Acute Coronary Events. Arch Intern Med. 2004 Jul 12;164(13):1457-63. doi: 10.1001/archinte.164.13.1457. PMID 15249356
- [Background] Steg PG, Iung B, Feldman LJ, Cokkinos D, Deckers J, Fox KA, Keil U, Maggioni AP. Impact of availability and use of coronary interventions on the prescription of aspirin and lipid lowering treatment after acute coronary syndromes. Heart. 2002 Jul;88(1):20-4. doi: 10.1136/heart.88.1.20. PMID 12067934
- [Background] Amar J, Chamontin B, Ferrieres J, Danchin N, Grenier O, Cantet C, Cambou JP. Hypertension control at hospital discharge after acute coronary event: influence on cardiovascular prognosis--the PREVENIR study. Heart. 2002 Dec;88(6):587-91. doi: 10.1136/heart.88.6.587. PMID 12433885
- [Background] Danchin N, Grenier O, Ferrieres J, Cantet C, Cambou JP. Use of secondary preventive drugs in patients with acute coronary syndromes treated medically or with coronary angioplasty: results from the nationwide French PREVENIR survey. Heart. 2002 Aug;88(2):159-62. doi: 10.1136/heart.88.2.159. PMID 12117845
- [Background] Zeller M, Cottin Y, Brindisi MC, Dentan G, Laurent Y, Janin-Manificat L, L'Huillier I, Beer JC, Touzery C, Makki H, Verges B, Wolf JE; RICO survey working group. Impaired fasting glucose and cardiogenic shock in patients with acute myocardial infarction. Eur Heart J. 2004 Feb;25(4):308-12. doi: 10.1016/j.ehj.2003.12.014. PMID 14984919
- [Background] Chambless L, Keil U, Dobson A, Mahonen M, Kuulasmaa K, Rajakangas AM, Lowel H, Tunstall-Pedoe H. Population versus clinical view of case fatality from acute coronary heart disease: results from the WHO MONICA Project 1985-1990. Multinational MONItoring of Trends and Determinants in CArdiovascular Disease. Circulation. 1997 Dec 2;96(11):3849-59. doi: 10.1161/01.cir.96.11.3849. PMID 9403607
- [Background] Marques-Vidal P, Ferrieres J, Metzger MH, Cambou JP, Filipiak B, Lowel H, Keil U. Trends in coronary heart disease morbidity and mortality and acute coronary care and case fatality from 1985-1989 in southern Germany and south-western France. Eur Heart J. 1997 May;18(5):816-21. doi: 10.1093/oxfordjournals.eurheartj.a015347. PMID 9152652
- [Result] Mesnier J, Cottin Y, Coste P, Ferrari E, Schiele F, Lemesle G, Thuaire C, Angoulvant D, Cayla G, Bouleti C, Gallet de Saint Aurin R, Goube P, Lhermusier T, Dillinger JG, Paganelli F, Saib A, Prunier F, Vanzetto G, Dubreuil O, Puymirat E, Boccara F, Eltchaninoff H, Cachanado M, Rousseau A, Drouet E, Steg PG, Simon T, Danchin N. Hospital admissions for acute myocardial infarction before and after lockdown according to regional prevalence of COVID-19 and patient profile in France: a registry study. Lancet Public Health. 2020 Oct;5(10):e536-e542. doi: 10.1016/S2468-2667(20)30188-2. Epub 2020 Sep 18. PMID 32950075
- [Derived] Gautier A, Danchin N, Ducrocq G, Rousseau A, Cottin Y, Cayla G, Prunier F, Durand-Zaleski I, Ravaud P, Angoulvant D, Coste P, Lemesle G, Bouleti C, Popovic B, Ferrari E, Silvain J, Dubreuil O, Lhermusier T, Goube P, Schiele F, Vanzetto G, Aboyans V, Gallet R, Eltchaninoff H, Thuaire C, Dillinger JG, Paganelli F, Gourmelen J, Steg PG, Simon T; FRENCHIE investigators. Rationale and design of the FRENch CoHort of myocardial Infarction Evaluation (FRENCHIE) study. Arch Cardiovasc Dis. 2024 Jun-Jul;117(6-7):417-426. doi: 10.1016/j.acvd.2024.04.004. Epub 2024 May 22. PMID 38821761